CLINICAL TRIAL: NCT00429195
Title: LIPGENE Dietary Intervention Study
Brief Title: The Effect of Dietary Fat Modification on Risk Factors Associated With the Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Collaborators: University of Reading (Other); University of Oslo (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Maastricht University Medical Center (Other); Universidad Nacional de Córdoba (Other); Jagiellonian University (Other); Uppsala University (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: LIPGENE Dietary Intervention
Record Dates: First submitted 2007-01-30; First posted 2007-01-31 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2007-01

CONDITIONS: Metabolic Syndrome
Keywords: LIPGENE; Fatty acid; Dietary intervention; Metabolic syndrome; Insulin resistance
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance

INTERVENTIONS:
Behavioral: Dietary Fatty Acid Modification

SUMMARY:
The LIPGENE Human Dietary Intervention Study, multi-centre, trans -European, single-blinded, randomised, controlled trial with two principal aims. Firstly to determine the relative efficacy of reducing dietary SFA consumption, by altering quality of dietary fat and reducing the quantity of dietary fat, on metabolic and molecular risk factors of the metabolic syndrome. Secondly to determine if common genetic polymorphisms affect an individual's responsiveness to dietary therapy.

DETAILED DESCRIPTION:
521 free-living subjects with the metabolic syndrome received one of four dietary treatments for 12 weeks: (1) High-fat (38% energy) SFA-rich diet; (2) High-fat (38% energy), MUFA-rich diet; (3) Isocaloric low-fat (28% energy), high-complex carbohydrate diet and (4) Isocaloric low-fat (28% energy), high-complex carbohydrate diet, with 1 g/d LC n-3 PUFA. A 3-day weighed food intake assessed dietary compliance pre-, mid- and post- intervention. An IVGTT, lipoprotein analysis, cytokine, adhesion molecule, coagulation factor and isoprostane levels were determined pre- and post-intervention. DNA, adipose and skeletal muscle biopsies, and PBMC were isolated to characterise nutrient sensitive molecular markers of insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Gender: males and females (not pregnant or lactating).
* Body Mass Index (BMI) 20-40 kg/m2
* Total cholesterol concentration equal to or < 8.0 mmol/l.
* Medications / nutritional supplements allowed, on condition that the subjects adhere to the same regimen during the intervention: anti-hypertensive medication (including beta-blockers), oral contraceptives, hormone replacement therapy, multi-vitamin supplements, other non-fatty acid based nutritional supplements (e.g. garlic, anti-oxidants, etc).
* Smokers and non-smokers.
* Regular consumers of alcohol, which is not excessive as defined by elevated liver enzymes (AST and ALT).
* Ethnicity: Intention to include white Europeans.

Exclusion Criteria:

* Diabetes or other endocrine disorders.
* Chronic inflammatory conditions.
* Kidney or liver dysfunction.
* Iron deficiency anaemia (haemoglobin < 12g/dl men, < 11g/dl women)
* Prescribed hypolipidaemic medication
* Prescribed anti-inflammatory medication
* Fatty acid supplements including fish oils, evening primrose oil, etc.
* Consumers of high doses of antioxidant vitamins (A, C, E, beta-carotene).
* Red rice yeast (Monascus purpureus) supplement usage.
* High consumers of oily fish (> 2 serving of oily fish per week of herring, mackerel, kippers, pilchards, sardines, salmon, trout, tuna (fresh), crabmeat or marlin). One portion is defined as a small herring or mackerel, one can of salmon or sardines or one salmon or tuna steak. Tinned tuna is permitted as it contains only minor amounts of long chain n-3 PUFAs.
* Highly trained or endurance athletes or those who participate in more than 3 periods of intense exercise per week.
* Volunteers planning to start a special diet or loose weight (e.g. the Slimfast Plan, Atkins Diet etc).
* Weight change equal or >3kg within the last 3 months.
* Alcohol or drug abuse (based on clinical judgement).
* Pregnant / lactating females / women planning a pregnancy in the next 12 months. Women who become pregnant during the dietary intervention period should be removed from the study.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480
Dates: Start 2004-02; Study Completion 2007-01

PRIMARY OUTCOMES:
IVGTT
Lipoprotein metabolism
Cytokine profiles
Coagulation
Fibrinolysis
Oxidative status

CONTACTS AND LOCATIONS:
Overall Officials: Helen M Roche, PhD, Study Director — University of Dublin, Trinity College; Christine Williams, PhD, Principal Investigator — University of Reading; Christian Drevon, MD, Principal Investigator — University of Oslo; Denis Larion, PhD, Principal Investigator — INSERM, Marseille; Wim Saris, PhD, Principal Investigator — Maastricht University; Jose Lopez Miranda, MD, PhD, Principal Investigator — Universidad de Córdoba; Aldona Dembinska-Kiec, MD, Principal Investigator — The Jagiellonian University Medical College; Bengt Vessby, MD, Principal Investigator — Uppsala University
Locations (1):
- Nutrigenomics Research Group, Institute of Molecular Medicine, University of Dublin, Trinity College, Dublin, Dublin, Ireland

REFERENCES:
- [Derived] Camargo A, Rangel-Zuniga OA, Alcala-Diaz J, Gomez-Delgado F, Delgado-Lista J, Garcia-Carpintero S, Marin C, Almaden Y, Yubero-Serrano EM, Lopez-Moreno J, Tinahones FJ, Perez-Martinez P, Roche HM, Lopez-Miranda J. Dietary fat may modulate adipose tissue homeostasis through the processes of autophagy and apoptosis. Eur J Nutr. 2017 Jun;56(4):1621-1628. doi: 10.1007/s00394-016-1208-y. Epub 2016 Mar 30. PMID 27029919
- [Derived] Yubero-Serrano EM, Delgado-Lista J, Tierney AC, Perez-Martinez P, Garcia-Rios A, Alcala-Diaz JF, Castano JP, Tinahones FJ, Drevon CA, Defoort C, Blaak EE, Dembinska-Kiec A, Riserus U, Lovegrove JA, Perez-Jimenez F, Roche HM, Lopez-Miranda J. Insulin resistance determines a differential response to changes in dietary fat modification on metabolic syndrome risk factors: the LIPGENE study. Am J Clin Nutr. 2015 Dec;102(6):1509-17. doi: 10.3945/ajcn.115.111286. Epub 2015 Nov 11. PMID 26561628
- [Derived] Delgado-Lista J, Perez-Martinez P, Solivera J, Garcia-Rios A, Perez-Caballero AI, Lovegrove JA, Drevon CA, Defoort C, Blaak EE, Dembinska-Kiec A, Riserus U, Herruzo-Gomez E, Camargo A, Ordovas JM, Roche H, Lopez-Miranda J. Top single nucleotide polymorphisms affecting carbohydrate metabolism in metabolic syndrome: from the LIPGENE study. J Clin Endocrinol Metab. 2014 Feb;99(2):E384-9. doi: 10.1210/jc.2013-3165. Epub 2013 Nov 7. PMID 24203067
- [Derived] Pena-Orihuela P, Camargo A, Rangel-Zuniga OA, Perez-Martinez P, Cruz-Teno C, Delgado-Lista J, Yubero-Serrano EM, Paniagua JA, Tinahones FJ, Malagon MM, Roche HM, Perez-Jimenez F, Lopez-Miranda J. Antioxidant system response is modified by dietary fat in adipose tissue of metabolic syndrome patients. J Nutr Biochem. 2013 Oct;24(10):1717-23. doi: 10.1016/j.jnutbio.2013.02.012. Epub 2013 May 3. PMID 23647888
- [Derived] Perez-Martinez P, Garcia-Rios A, Delgado-Lista J, Gjelstad IM, Gibney J, Kiec-Wilk B, Camargo A, Helal O, Karlstrom B, Blaak EE, Hall W, Riserus U, Dembinska-Kiec A, Defoort C, Saris WH, Lovegrove JA, Drevon CA, Roche HM, Lopez-Miranda J. Gene-nutrient interactions on the phosphoenolpyruvate carboxykinase influence insulin sensitivity in metabolic syndrome subjects. Clin Nutr. 2013 Aug;32(4):630-5. doi: 10.1016/j.clnu.2012.10.003. Epub 2012 Oct 8. PMID 23092637
- [Derived] Camargo A, Rangel-Zuniga OA, Pena-Orihuela P, Marin C, Perez-Martinez P, Delgado-Lista J, Gutierrez-Mariscal FM, Malagon MM, Roche HM, Tinahones FJ, Perez-Jimenez F, Lopez-Miranda J. Postprandial changes in the proteome are modulated by dietary fat in patients with metabolic syndrome. J Nutr Biochem. 2013 Jan;24(1):318-24. doi: 10.1016/j.jnutbio.2012.06.014. Epub 2012 Sep 5. PMID 22959058
- [Derived] Perez-Martinez P, Perez-Caballero AI, Garcia-Rios A, Yubero-Serrano EM, Camargo A, Gomez-Luna MJ, Marin C, Gomez-Luna P, Dembinska-Kiec A, Rodriguez-Cantalejo F, Tinahones FJ, Roche HM, Perez-Jimenez F, Lopez-Miranda J, Delgado-Lista J. Effects of rs7903146 variation in the Tcf7l2 gene in the lipid metabolism of three different populations. PLoS One. 2012;7(8):e43390. doi: 10.1371/journal.pone.0043390. Epub 2012 Aug 20. PMID 22916254
- [Derived] van Hees AM, Jocken JW, Essers Y, Roche HM, Saris WH, Blaak EE. Adipose triglyceride lipase and hormone-sensitive lipase protein expression in subcutaneous adipose tissue is decreased after an isoenergetic low-fat high-complex carbohydrate diet in the metabolic syndrome. Metabolism. 2012 Oct;61(10):1404-12. doi: 10.1016/j.metabol.2012.03.017. Epub 2012 Apr 30. PMID 22551950
- [Derived] Delgado-Lista J, Perez-Martinez P, Garcia-Rios A, Phillips CM, Hall W, Gjelstad IM, Lairon D, Saris W, Kiec-Wilk B, Karlstrom B, Drevon CA, Defoort C, Blaak EE, Dembinska-Kiec A, Riserus U, Lovegrove JA, Roche HM, Lopez-Miranda J. A gene variation (rs12691) in the CCAT/enhancer binding protein alpha modulates glucose metabolism in metabolic syndrome. Nutr Metab Cardiovasc Dis. 2013 May;23(5):417-23. doi: 10.1016/j.numecd.2011.09.008. Epub 2012 Jan 23. PMID 22269963
- [Derived] Paniagua JA, Perez-Martinez P, Gjelstad IM, Tierney AC, Delgado-Lista J, Defoort C, Blaak EE, Riserus U, Drevon CA, Kiec-Wilk B, Lovegrove JA, Roche HM, Lopez-Miranda J; LIPGENE Study Investigators. A low-fat high-carbohydrate diet supplemented with long-chain n-3 PUFA reduces the risk of the metabolic syndrome. Atherosclerosis. 2011 Oct;218(2):443-50. doi: 10.1016/j.atherosclerosis.2011.07.003. Epub 2011 Jul 12. PMID 21839455
- [Derived] Jans A, Sparks LM, van Hees AM, Gjelstad IM, Tierney AC, Riserus U, Drevon CA, Roche HM, Schrauwen P, Blaak EE. Transcriptional metabolic inflexibility in skeletal muscle among individuals with increasing insulin resistance. Obesity (Silver Spring). 2011 Nov;19(11):2158-66. doi: 10.1038/oby.2011.149. Epub 2011 Jun 23. PMID 21701566
- [Derived] Perez-Martinez P, Delgado-Lista J, Garcia-Rios A, Mc Monagle J, Gulseth HL, Ordovas JM, Shaw DI, Karlstrom B, Kiec-Wilk B, Blaak EE, Helal O, Malczewska-Malec M, Defoort C, Riserus U, Saris WH, Lovegrove JA, Drevon CA, Roche HM, Lopez-Miranda J. Glucokinase regulatory protein genetic variant interacts with omega-3 PUFA to influence insulin resistance and inflammation in metabolic syndrome. PLoS One. 2011;6(6):e20555. doi: 10.1371/journal.pone.0020555. Epub 2011 Jun 6. PMID 21674002
- [Derived] Perez-Martinez P, Delgado-Lista J, Garcia-Rios A, Ferguson JF, Gulseth HL, Williams CM, Karlstrom B, Kiec-Wilk B, Blaak EE, Helal O, Malczewska-Malec M, Defoort C, Riserus U, Saris WH, Lovegrove JA, Drevon CA, Roche HM, Lopez-Miranda J. Calpain-10 interacts with plasma saturated fatty acid concentrations to influence insulin resistance in individuals with the metabolic syndrome. Am J Clin Nutr. 2011 May;93(5):1136-41. doi: 10.3945/ajcn.110.010512. Epub 2011 Mar 9. PMID 21389182
- [Derived] Jimenez-Gomez Y, Marin C, Peerez-Martinez P, Hartwich J, Malczewska-Malec M, Golabek I, Kiec-Wilk B, Cruz-Teno C, Rodriguez F, Gomez P, Gomez-Luna MJ, Defoort C, Gibney MJ, Perez-Jimenez F, Roche HM, Lopez-Miranda J. A low-fat, high-complex carbohydrate diet supplemented with long-chain (n-3) fatty acids alters the postprandial lipoprotein profile in patients with metabolic syndrome. J Nutr. 2010 Sep;140(9):1595-601. doi: 10.3945/jn.109.120816. Epub 2010 Jul 14. PMID 20631323
- [Derived] Ferguson JF, Phillips CM, McMonagle J, Perez-Martinez P, Shaw DI, Lovegrove JA, Helal O, Defoort C, Gjelstad IM, Drevon CA, Blaak EE, Saris WH, Leszczynska-Golabek I, Kiec-Wilk B, Riserus U, Karlstrom B, Lopez-Miranda J, Roche HM. NOS3 gene polymorphisms are associated with risk markers of cardiovascular disease, and interact with omega-3 polyunsaturated fatty acids. Atherosclerosis. 2010 Aug;211(2):539-44. doi: 10.1016/j.atherosclerosis.2010.03.027. Epub 2010 Mar 27. PMID 20409549
- [Derived] van Hees AM, Saris WH, Hul GB, Schaper NC, Timmerman BE, Lovegrove JA, Roche HM, Blaak EE. Effects of dietary fat modification on skeletal muscle fatty acid handling in the metabolic syndrome. Int J Obes (Lond). 2010 May;34(5):859-70. doi: 10.1038/ijo.2010.6. Epub 2010 Feb 2. PMID 20125104
- [Derived] Ferguson JF, Phillips CM, Tierney AC, Perez-Martinez P, Defoort C, Helal O, Lairon D, Planells R, Shaw DI, Lovegrove JA, Gjelstad IM, Drevon CA, Blaak EE, Saris WH, Leszczynska-Golabek I, Kiec-Wilk B, Riserus U, Karlstrom B, Miranda JL, Roche HM. Gene-nutrient interactions in the metabolic syndrome: single nucleotide polymorphisms in ADIPOQ and ADIPOR1 interact with plasma saturated fatty acids to modulate insulin resistance. Am J Clin Nutr. 2010 Mar;91(3):794-801. doi: 10.3945/ajcn.2009.28255. Epub 2009 Dec 23. PMID 20032495
- [Derived] Hartwich J, Malec MM, Partyka L, Perez-Martinez P, Marin C, Lopez-Miranda J, Tierney AC, Mc Monagle J, Roche HM, Defoort C, Wolkow P, Dembinska-Kiec A. The effect of the plasma n-3/n-6 polyunsaturated fatty acid ratio on the dietary LDL phenotype transformation - insights from the LIPGENE study. Clin Nutr. 2009 Oct;28(5):510-5. doi: 10.1016/j.clnu.2009.04.016. Epub 2009 May 28. PMID 19481310